CLINICAL TRIAL: NCT05504655
Title: Safety and Efficacy of N-Acetylcysteine as an Adjuvant Therapy in Critically Ill COVID-19 Patients: A Retrospective Observational Study
Brief Title: N-Acetylcysteine as an Adjuvant Therapy in Critically Ill COVID-19 Patients:
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hanaa Mohamed Abdallah ElGendy MD, Professor, Ain Shams University
Other Study IDs: FMASU 129/2022. FWA 000017585
Record Dates: First submitted 2022-08-13; First posted 2022-08-17 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational NAC group: Based on a FDA approved 3-bag regime, NAC (Molecular weight:163) was administrated intravenously, initially 150 mg/kg in 200 mL of 0.9%NaCL for 60 minutes (first bag), followed by 50 mg/kg in 500 mL of 0.9%NaCL for 4 hours (second bag), and then 100 mg/kg in 1000 mL of 0.9%NaCL for 16 hours (third bag)
- Observational Non NAC group: N-acetylcysteine given IV at 600 mg every 12 hours till discharge from ICU.

SUMMARY:
In this study, we retrospectively will investigate safety and efficacy of NAC dose given in paracetamol toxicity as an adjuvant therapy in critically ill COVID-19 patients with acute respiratory distress and determine whether NAC in high doses can avoid respiratory failure in patients with COVID-19.

DETAILED DESCRIPTION:
Type of Study:Retrospective Observational Cohort Study. Study Setting: Ain shams university hospitals . Study Period: from December 2020 to February 2022 Study Population:Patients aged 18 years or older of both genders diagnosed with confirmed critically ill COVID-19 .

This is a retrospective observational study in which all cases will be collected from ICU of Ain shams university hospitals during COVID-19 outbreak. All data will be extracted from clinical records. All patients initially admitted to ICU with SPO2 less than 94 % will be included between December 2020 to February 2022. Infection with COVID-19 was confirmed by PCR. All patients received standard care, according to the institutional protocol.

Laboratory and Radiological Investigations Demographic, clinical, laboratory, management, and outcome data will be obtained from the medical records. Routine laboratory tests were done for all patients, including CBC, C-reactive protein, renal profile, coagulation profile, liver profile, lactate, electrolytes, procalcitonin, ferritin and D-dimer.Infection with COVID-19 was confirmed by reverse transcriptase-polymerase chain reaction (RT-PCR) assay of nasopharyngeal swab. Chest computed tomography (CT) was also done for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Oxyhemoglobin saturation (SaO2) of less than 94% while breathing ambient air

Exclusion Criteria:

* Need for immediate mechanical ventilation on admission, known allergy or hypersensitivity to NAC, end stage renal and liver diseases, heart failure and pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older of both genders diagnosed with confirmed critically ill COVID-19
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
The necessity for invasive mechanical ventilation | 3 to 4 months
  Primary outcome

SECONDARY OUTCOMES:
The onset and duration of invasive mechanical ventilation, length of ICU stay, length of hospital stay and 28 days mortality | 3 to 4 months
  Secondary outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Hanaa El Gendy, Cairo, Ain Shams University Specialized Hospital, Egypt

IPD SHARING:
Plan to Share IPD: No